CLINICAL TRIAL: NCT02928978
Title: TBCRC 042 - A Randomized Phase II Window-of-Opportunity Trial of Ruxolitinib in Patients With High Risk and Premalignant Breast Conditions
Brief Title: Ruxolitinib for Premalignant Breast Disease
Acronym: TBCRC042
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Julie Nangia (Other)
Collaborators: Incyte Corporation (Industry); Translational Breast Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Julie Nangia, Assistant Professor, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-38855
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Ductal Carcinoma In Situ; Atypical Lobular Hyperplasia; Atypical Ductal Hyperplasia; Lobular Carcinoma In Situ
Keywords: Premalignant Breast Disease; ALH; ADH; DCIS; LCIS; Breast Cancer Prevention; Ruxolitinib
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ruxolitinib (Experimental): Participants will receive ruxolitinib 20 mg by mouth twice daily for 15 days (+/- 5 days). Ruxolitinib will be supplied as four, 5 mg tablets.
  Interventions: Drug: Ruxolitinib
- Placebo (Placebo Comparator): Participants will receive a placebo (sugar pill) that is designed to mimic ruxolitinib. The placebo will be supplied as four, 5 mg tablets. Participants assigned to this arm will take four, 5 mg tablets by mouth twice daily for 15 days (+/- 5 days).
  Interventions: Drug: Placebo (for Ruxolitinib)

INTERVENTIONS:
Drug: Ruxolitinib — tablet (taken by mouth)
  Other Names: Jakafi; INCB018424
  Arms: Ruxolitinib
Drug: Placebo (for Ruxolitinib) — tablet (taken by mouth)
  Arms: Placebo

SUMMARY:
This study is evaluating how ruxolitinib affects premalignant breast cells. One half of the study participants will receive ruxolitinib for approximately 15 days, and the other half will receive a placebo (sugar pill) for approximately 15 days. Once study participants have completed their ruxolitinib or placebo, participants will undergo surgery to remove the premalignant breast tissue.

ELIGIBILITY:
Inclusion Criteria:

* Have a breast biopsy showing ADH (atypical ductal hyperplasia), ALH (atypical lobular hyperplasia), LCIS (lobular carcinoma in situ), or DCIS (ductal carcinoma in situ) requiring surgical excision. Microinvasive disease is allowed.

  * NOTE: Tissue from the diagnostic biopsy must be accessible/available for research correlates (i.e., a tissue block or ~10 unstained slides). Due to the nature of the study, fewer slides may be accepted with prior permission from the Protocol Chair if there is insufficient tissue.
* Women and men age 18 and older.
* Adequate hematologic and organ function, defined as follows:

  * Absolute neutrophil count ≥ 1500/mm3
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet levels >200 x 109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
  * AST/ALT ≤ 2.5 x institutional ULN
  * Alkaline phosphatase ≤ 5 x institutional ULN
  * Creatinine clearance > 50 mL/min as calculated by the Cockcroft-Gault method
* Willing to not use concomitant strong CYP3A4 inhibitors as this could interfere with the metabolism of ruxolitinib (i.e azole antifungals, clarithromycin, conivaptan, grapefruit juice, mibefradil, nefazodone, protease inhibitors, telithromycin).
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* If the patient undergoes germline genetic testing, the results must be received prior to randomization, as the results may affect the surgical approach and, in turn, the date of surgical excision.
* Patient understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign a written informed consent document.

Exclusion Criteria:

* Treatment with selective estrogen receptor modulators (SERMs) or aromatase inhibitors for breast cancer prevention within 1 year prior to starting study treatment.
* Treatment with any other investigational agents within 30 days of starting study treatment.
* Current diagnosis of invasive breast cancer (current microinvasive disease is allowed), or previous history of invasive breast cancer diagnosed within the last 5 years.

NOTE: If previous history of ER+ invasive breast cancer diagnosed > 5 years ago, patient must be off endocrine therapy for at least 1 year prior to starting study treatment.

* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, end stage renal disease (ESRD), or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or nursing.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ruxolitinib.
* Prior or current treatment with a JAK inhibitor, for any indication.
* Known active Hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Apoptosis | 15 days (+/- 5 days)
  The number of premalignant breast cells in apoptosis at the time of diagnosis will be compared to the number of cells in apoptosis following treatment with 15 (+/- 5) days of ruxolitinib or placebo.

SECONDARY OUTCOMES:
pSTAT5 | 15 days (+/- 5 days)
  To determine the difference in change in pSTAT5 levels between diagnosis and surgery as a function of ruxolitinib treatment versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Julie Nangia, M.D., Principal Investigator — Baylor College of Medicine
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas
  - O'Quinn Medical Tower - McNair Campus; Dan L Duncan Comprehensive Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No